CLINICAL TRIAL: NCT02096003
Title: Comparison of Intrathecal Hydromorphone and Intrathecal Morphine for Postoperative Analgesia After Cesarean Delivery
Brief Title: Intrathecal Hydromorphone for Pain Control After Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Yaakov Beilin, Professor of Anesthesiology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 13-1762
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Pain; Cesarean Section
Keywords: Intrathecal hydromorphone; Intrathecal morphine; Primary cesarean section; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal morphine (Active Comparator): 0.25mg ( 250mcg) intrathecal morphine added to 1.5 mg 0.75% bupivicaine for single shot spinal anesthesia in primary cesarean sections
  Interventions: Drug: Intrathecal morphine
- Intrathecal hydromorphone (Experimental): 50mcg intrathecal hydromorphone added to 1.5 mg 0.75% bupivicaine for single shot spinal anesthesia in primary cesarean sections.
  Interventions: Drug: Intrathecal hydromorphone

INTERVENTIONS:
Drug: Intrathecal morphine — 0.25mg intrathecal morphine is the standard opioid medication the investigators use for analgesia for cesarean sections. It is the control arm.
  Other Names: Duramorph
  Arms: Intrathecal morphine
Drug: Intrathecal hydromorphone — 50mcg intrathecal hydromorphone will be added to 1.5mg 0.75% bupivicaine for single shot spinal anesthesia.
  Other Names: Dilaudid
  Arms: Intrathecal hydromorphone

SUMMARY:
The use of intrathecal opioids for analgesia in the setting of cesarean section has become standard obstetric anesthesia practice. Currently, two opioids are commonly used. These opioids are fentanyl and morphine (Duramorph). Intrathecal opioids are an excellent source of analgesia and act to reduce the stress response to surgery.

Currently, most obstetric anesthesiologists use intrathecal morphine for analgesia after cesarean delivery. Morphine provides excellent analgesia for cesarean section. However, use of this medication is associated with side effects such as pruritus and nausea and vomiting.

Recently, multiple obstetric anesthesia groups began to use intrathecal hydromorphone for cesarean delivery when morphine was unavailable. As groups began to use hydromorphone, retrospective data became available that demonstrated its safety and efficacy for use during cesarean section.

In order to fully elucidate the analgesic and side effect properties of hydromorphone for cesarean delivery, a prospective randomized, double blind study comparing morphine and hydromorphone is necessary. The investigators need to understand whether hydromorphone is as effective as morphine for analgesia after cesarean section, and whether it is associated with fewer or more side effects. The results of the study will allow providers to make educated decisions to better care for their patient.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary cesarean section
* Females age 18-40

Exclusion Criteria:

* Emergency cesarean section
* Anesthetic other than spinal
* History of chronic pain or pre-op opioid use
* Allergy to morphine or hydromorphone
* BMI>40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Beilin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in April 2014 with enrollment from May 2014 to May 2017
Period: Overall Study
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
Started | 40 | 40
Completed | 38 | 37
Not Completed | 2 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — additional surgery | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (5.1) | 33.75 (4.1) | 34.1 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Fentanyl PCA Consumption
Description: Total dose of fentanyl patient controlled analgesia (pca) used in 24 hours post-op.
Time Frame: at 24 hours
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
Number analyzed (Participants) | 38 | 37
µg | 300 (432) | 446 (440)

2. Secondary Outcome: Time to Initial PCA Use
Description: When does the patient need to use the PCA for the first time? This will be used to assess when morphine and hydromorphone first begin to provide analgesia.
Time Frame: up to 24 hours
Population: data not collected.
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pain Score
Description: Assess pain scores on a scale of 1-5, with higher score indicating more pain.
Time Frame: at 24 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
Number analyzed (Participants) | 38 | 37
score on a scale | 4.8 [1 to 5] | 4.7 [1 to 5]

4. Secondary Outcome: Patient Satisfaction Score
Description: Patient satisfaction score - total scale of 1-5, with higher score indicating more satisfaction
Time Frame: at 24 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
Number analyzed (Participants) | 38 | 37
score on a scale | 4.8 [1 to 5] | 4.6 [1 to 5]

5. Secondary Outcome: Symptom Scale for Two Specific Side Effects of Nausea and Pruritus
Description: Symptom scale for nausea and pruritus. Full scale from 1-5, with higher score indicating more symptoms.
Time Frame: up to 24 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
Number analyzed (Participants) | 38 | 37
score on a scale
  Nausea | 4.4 [1 to 5] | 4.7 [1 to 5]
  Pruritus | 3.8 [1 to 5] | 4 [1 to 5]

ADVERSE EVENTS:
Time Frame: up to 24 hours
Arm/Group | Intrathecal Morphine | Intrathecal Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 36/40 | 35/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intrathecal Morphine (N=40) | Intrathecal Hydromorphone (N=40)
Nausea (General disorders) | 2 | 3
Puritus (Skin and subcutaneous tissue disorders) | 34 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT02096003/Prot_SAP_000.pdf